CLINICAL TRIAL: NCT06731296
Title: Characteristics of General Surgery Patients Admitted to the Intensive Care Unit, Villavicencio, 2022-2024.
Brief Title: General Surgery Patients at the Intensive Care Unit
Acronym: TraViII
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Departamental de Villavicencio (Other)
Responsible Party: Principal Investigator, Norton Perez-Gutierrez, MD, ICU chief of staff, Hospital Departamental de Villavicencio
Other Study IDs: GRIVI_2024_01_QX_UCI
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Critical Illness; Postoperative Complications
Keywords: Acute Care Surgery; Operative Surgical Procedures; Perioperative Care; Critical Care; Intensive Care Units; In-hospital Mortality; Colombia
MeSH Terms: conditions — Critical Illness; Postoperative Complications

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Abdominal surgery: Patients admitted to the ICU after an abdominal surgery.
  Interventions: Other: Presence of a risk factor
- Older adults: Older adults (65+) surgical patients admitted to the ICU.
  Interventions: Other: Presence of a risk factor

INTERVENTIONS:
Other: Presence of a risk factor — Demographic, severity, type of surgery, diagnosis, diagnostic system, type of admission.

SUMMARY:
Introduction: high-risk surgical patients in the intensive care unit (ICU) are a unique population that has yet to be carefully monitored. Unlike most publications, which focus on general ICU patients, this study aims to fill a gap by specifically evaluating factors associated with lethal outcomes for surgical patients in the ICU.

Methodology: An analytical cross-sectional trial was designed to answer the research question and be performed it in one or two institutions with a median and high complexity of care in the Orinoco region. ICU discharge book registries will be selected from a post-pandemic period (2022-2024). Adult and pediatric patients admitted from the surgical theatre by emergency or elective surgical procedures or with ICD-10 (International Classification of Diseases 10th revision) codes related to the pediatric or general surgery specialty. The frequency and proportion of categorical variables and the central distribution and dispersion of quantitative variables will be described. Chi-square and U-Mann & Whitney tests will be used to compare variables. A p-value <0.05 will be selected as statistical significance.

Results: The researchers expect to find the demographic characteristics of surgical patients admitted to the ICU by diagnostic groups and by severity associated with mortality.

Conclusions: The trial, which is both feasible and necessary, has the potential to provide valuable insights into the factors affecting outcomes for high-risk surgical patients at the ICU. This knowledge could lead to improved patient care and outcomes, making the research essential and highly beneficial.

DETAILED DESCRIPTION:
Introduction: high-risk surgical patients in the intensive care unit (ICU) are a unique population that has yet to be carefully monitored to minimize surgical or non-surgical complications. It is necessary to identify factors associated with adverse outcomes. Unlike most publications, which focus on general ICU patients, this study aims to fill a gap by specifically evaluating factors associated with lethal outcomes for surgical patients in the ICU.

Methodology: An analytical cross-sectional trial was designed to answer the research question and be performed it in one or two institutions with a median and high complexity of care in the Orinoco region. ICU discharge book registries will be selected from a post-pandemic period (2022-2024). Adult and pediatric patients admitted from the surgical theatre by emergency or elective surgical procedures or with ICD-10 (International Classification of Diseases 10th revision) codes related to the pediatric or general surgery specialty. The frequency and proportion of categorical variables and the central distribution and dispersion of quantitative variables will be described. Chi-square and U-Mann & Whitney tests will be used to compare variables. A p-value <0.05 will be selected as statistical significance.

Results: The researchers expect to find the demographic characteristics of surgical patients admitted to the ICU by diagnostic groups and by severity associated with mortality to establish predictive models of adverse outcomes in the admission to the intensive care unit to implement early preventive interventions.

Conclusions: The trial, which is both feasible and necessary, has the potential to provide valuable insights into the factors affecting outcomes for high-risk surgical patients at the ICU. This knowledge could lead to improved patient care and outcomes, making the research essential and highly beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a surgical diagnosis admitted to the ICU.
* Patients in the operative period admitted to the ICU.

Exclusion Criteria:

* Patients admitted from another hospital.
* Surgical procedures performed in another hospital.
* Surgical patients referred to another hospital.

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General surgery patients admitted to the ICU, especially for postoperative care.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | 30 days
  ICU discharges due to patient death in the ICU.

SECONDARY OUTCOMES:
ICU length of stay | 30 days
  ICU length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Norton Perez, MD, Principal Investigator — Universidad Cooperativa de Colombia; Hospital Departamental de Villavicencio; Clínica Primavera
Locations (2):
- Colombia (2):
  - Clinica Primavera, Villavicencio, Meta Department
  - Hospital Departamental de Villavicencio, Villavicencio, Meta Department

IPD SHARING:
Plan to Share IPD: No
The data contains sensitive information of patients.

REFERENCES:
- [Result] Dovzhanskiy DI, Schwab S, Bischoff MS, Brenner T, Weigand MA, Hinz U, Bockler D. Extended intensive care correlates with worsening of surgical outcome after elective abdominal aortic reconstruction. J Cardiovasc Surg (Torino). 2021 Dec;62(6):591-599. doi: 10.23736/S0021-9509.21.11842-7. Epub 2021 May 20. PMID 34014060
- [Result] Menzenbach J, Layer YC, Layer YL, Mayr A, Coburn M, Wittmann M, Hilbert T. The level of postoperative care influences mortality prediction by the POSPOM score: A retrospective cohort analysis. PLoS One. 2021 Sep 29;16(9):e0257829. doi: 10.1371/journal.pone.0257829. eCollection 2021. PMID 34587207
- [Result] Hynes AM, Lambe LD, Scantling DR, Bormann BC, Atkins JH, Rassekh CH, Seamon MJ, Martin ND. A surgical needs assessment for airway rapid responses: A retrospective observational study. J Trauma Acute Care Surg. 2022 Jan 1;92(1):126-134. doi: 10.1097/TA.0000000000003348. PMID 34252060
- [Result] Peters F, Hohenstein S, Bollmann A, Kuhlen R, Ritz JP. The Postoperative Utilization of Intensive Care Beds After Visceral Surgery Procedures. Dtsch Arztebl Int. 2023 Sep 22;120(38):633-638. doi: 10.3238/arztebl.m2023.0158. PMID 37427992
- [Result] Timan TJ, Karlsson O, Sernert N, Prytz M. Standardized perioperative management in acute abdominal surgery: Swedish SMASH controlled study. Br J Surg. 2023 May 16;110(6):710-716. doi: 10.1093/bjs/znad081. PMID 37071812
- [Result] Chinawong C, Utriyaprasit K, Sindhu S, Viwatwongkasem C, Suksompong S. Factors Influencing Pre-Cardiopulmonary Arrest Signs among Post-General Surgery Patients in Critical Care Service System. Int J Environ Res Public Health. 2023 Jan 3;20(1):876. doi: 10.3390/ijerph20010876. PMID 36613197
- [Result] Meschino MT, Vogt KN, Allen L, Saddik M, Nenshi R, Van Heest R, Saleh F, Widder S, Minor S, Joos E, Parry NG, Murphy PB, Ball CG, Hameed M, Engels PT; CANUCS (Canadian Collaborative on Urgent Care Surgery). Operating room use for emergency general surgery cases: analysis of the Patterns of Complex Emergency General Surgery in Canada study. Can J Surg. 2023 Jan 3;66(1):E13-E20. doi: 10.1503/cjs.008120. Print 2023 Jan-Feb. PMID 36596587
- [Result] Suarez-de-la-Rica A, Ripolles-Melchor J, Aldecoa C, Abad-Motos A, Ferrando C, Abad-Gurumeta A, Diaz-Almiron M, Gil-Lapetra C, Garcia-Miguel FJ, Pedregosa-Sanz A, Esteve-Perez N, Rodriguez-Jimenez R, Gimeno Fernandez P, Maseda E; POWER Study Investigators Group for the Spanish Perioperative Audit and Research Network (RedGERM-SPARN). Postoperative Critical Care Admission Was Not Associated with Improved Postoperative Outcomes in Elective Colorectal Surgery: Secondary Analysis Of POWER Trial. J Gastrointest Surg. 2023 Oct;27(10):2187-2198. doi: 10.1007/s11605-023-05780-z. Epub 2023 Aug 7. PMID 37550589
- [Result] Yohann A, Kayange L, Purcell L, Gallaher J, Charles A. Acute care surgery in a Malawian district hospital: Epidemiology, outcomes, and assessment of operative capacity. Trop Doct. 2023 Jan;53(1):73-80. doi: 10.1177/00494755221102226. Epub 2022 Jul 27. PMID 35895502
- [Result] Stahlschmidt A, Passos SC, Cardoso GR, Schuh GJ, Neto PCDS, Castro SMJ, Stefani LC. Postoperative intensive care allocation and mortality in high-risk surgical patients: evidence from a low- and middle-income country cohort. Braz J Anesthesiol. 2024 Jul-Aug;74(4):844517. doi: 10.1016/j.bjane.2024.844517. Epub 2024 May 23. PMID 38789003